CLINICAL TRIAL: NCT01211041
Title: The Relationship Between Morphology and Virulent Genes of Candida Albicans and Clinical Aspects, Surveillance of Fungemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Tsong-Yih Ou, Infectious Disease Department
Other Study IDs: 99026
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Candidemia Prognostic Factor and Mycobiological Analysis.
Keywords: Candida albicans, fungemia , prognostic factor
MeSH Terms: conditions — Fungemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Candida albicans is the most common and important clinical fungal pathogen. Our previous surveillance disclosed that fluconazole could induce different morphological changes in clinical strains. Our current study on C. albicans causing candiuria disclosed that renal insufficiency , diabetes mellitus, respiratory failure and uremia were risk factors of treatment failure. However, we also found results of E-test drug susceptible test could not predict outcome. Hence, retrospective analysis of 31 months period, cases that had C. albicans inducing candidemia were reviewed and 60 cases were enrolled for morphological study and potential virulent gene analysis.

This study is designed to clarity the clinical meaning of morphological form and virulent genes on candidemia. To do this study is probably helpful for treatment of candidiasis.

ELIGIBILITY:
Inclusion Criteria:

* 2007 to 2010 medical records
* Cases with candidemmia of Candida albicans with available clinical information in medical records for analysis.
* Cases with candidemmia of Candida albicans which clinical isolates were preserved.

Exclusion Criteria:

* Cases were not hospitalized for treatment and data were not available for analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: case with candidemia of Candida albicans and candida caused the disease .
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tsong-Yih Ou, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan